CLINICAL TRIAL: NCT05094505
Title: Isolated and Combined Effect of a Low Carbohydrate Diet and Chronic Exercise Exposure to Hypoxia on Glycaemic Control and Cardiovascular Risk Factors in Patients With Type 2 Diabetes
Brief Title: Isolated and Combined Effect of a Low Carbohydrate Diet and Exercise in Hypoxia in Patients With Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade do Porto (Other)
Collaborators: Fundação para a Ciência e a Tecnologia (Other); University Institute of Maia (Other)
Responsible Party: Principal Investigator, Raquel Kindlovits, PhD student, Universidade do Porto
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BD2020.06520
Record Dates: First submitted 2021-09-15; First posted 2021-10-26 (Actual); Last update posted 2023-07-19 (Actual); Status verified 2023-07

CONDITIONS: Carbohydrate; Hypoxia; Exercise; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Hypoxia; Motor Activity; Diabetes Mellitus, Type 2 | interventions — Exercise; Diet, Carbohydrate-Restricted

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- CONTROL GROUP (Active Comparator): Exercise at sea level, normoxia. Control diet.
  Interventions: Other: Exercise in normoxia; Other: Control diet
- Ex. Hyp. GROUP (Experimental): Exercise in hypoxia at 3000m altitude. Control diet.
  Interventions: Other: Control diet; Other: Exercise in hypoxia
- Ex. Hyp. + LCD GROUP (Experimental): Exercise in hypoxia at 3000m altitude. Low carbohydrate diet.
  Interventions: Other: Exercise in hypoxia; Other: Low carbohydrate diet

INTERVENTIONS:
Other: Exercise in normoxia — Exercise at sea level, 3 sessions per week, during a 8-week period intervention and will consist in 60 min on an ergometer, of continuous moderate and high intensity interval training. . All exercise testing and training sessions will be carried out at the same time of day (± 2 hours) and visits will be separated by at least 48h of recovery.
  Arms: CONTROL GROUP
Other: Control diet — Control diet: diet plans will be individualized and energy-content prescriptions will be constant throughout the study to maintain the isocaloric control between diets. The planned macronutrient compositions will be 20% of energy from fat, 20% from protein and 60% from carbohydrates for the low-fat diet during the 8 weeks. Diets emphasis on low-glycemic index foods and limited saturated fat to 10% of energy. Participants will meet individually with a dietitian two times for 8 weeks and should start the dietary intervention along with the intervention with exercise.
  Arms: CONTROL GROUP; Ex. Hyp. GROUP
Other: Exercise in hypoxia — Exercise at 3000m altitude, 3 sessions per week, during a 8-week period intervention and will consist in 60 min on an ergometer, of continuous moderate and high intensity interval training. . All exercise testing and training sessions will be carried out at the same time of day (± 2 hours) and visits will be separated by at least 48h of recovery.
  Arms: Ex. Hyp. + LCD GROUP; Ex. Hyp. GROUP
Other: Low carbohydrate diet — Low carbohydrate diet: diet plans will be individualized and energy-content prescriptions will be constant throughout the study to maintain the isocaloric control between diets. The planned macronutrient compositions will be 40% of energy from fat, 20% from protein and 40% from carbohydrates for the low-fat diet during the 8 weeks. Diets emphasis on low-glycemic index foods and limited saturated fat to 10% of energy. Participants will meet individually with a dietitian two times for 8 weeks and should start the dietary intervention along with the intervention with exercise.
  Arms: Ex. Hyp. + LCD GROUP

SUMMARY:
The purpose of this study is to determine the effects of isolated chronic exercise in hypoxia and combined exercise in hypoxia with a low carbohydrate diet on hypoxia-induced transcription factor (HIF1-α); glycaemic control and cardiovascular risk factors in patients with type 2 diabetes.

DETAILED DESCRIPTION:
At baseline, diet plans will be individualized and energy-content prescriptions will be constant throughout the study to maintain the isocaloric control between diets. The planned macronutrient compositions will be, 30% of energy from carbohydrates, 20% from protein and 50% from fat for low carbohydrate diet (LCD) and 30% of energy from fat, 20% from protein and 50% from carbohydrates for the low-fat diet (control diet), during the 8 weeks. Both diets emphasis on low-glycemic index foods and limited saturated fat to 10% of energy, and calculated with appropriate software.

Exercise in hypoxia (at 3000m altitude, 3 sessions/week) will occur during a 8-week period intervention and all testing sessions carried out in a hypoxic chamber at Exercise Medical Center, Porto - Portugal. This chamber allows control of O2 (11-20.97%), temperature (until 50ºC), humidity (until 80%) and altitude (until 8000m). Exercise in hypoxia sessions will consist in 60 min on an ergometer (Excalibur, Lode, Netherlands) of continuous moderate and high intensity interval training, these latter considered as an efficient strategy to improve cardiorespiratory and metabolic health in patients with type 2 diabetes. Loads will be quantified according to pre-intervention testing assessments and controlled throughout each training session. All exercise testing and training sessions will be carried out at the same time of day (± 2 hours) and visits will be separated by at least 48h of recovery.

Height will be measured with use of a stadiometer (SECA), waist circumference was measured by using a tape measure positioned 3 cm above the iliac crest. Body mass index (BMI), weight, fat mass (FM) and fat-free mass (FFM) were determined by using whole-body dual-energy X-ray absorptiometry (Lunar Prodigy; General Electric Corp.). Blood pressure will be measured by using an automated sphygmomanometer (Dinamap Pro; Medical Systems,Tampa, FL) and haematological adaptations will be measured by collecting a venous blood sample from a vein in the arm using a needle. A total of 3 blood samples (pre, 1h post first intervention testing and 48h post the last intervention testing) will be taken.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of type 2 diabetes for at least one year
* Glycosylated haemoglobin less than 10%
* Pharmacological regimen stabilized for at least three months
* Main complications of diabetes tracked and controlled (diabetic retinopathy, diabetic nephropathy, diabetic foot and main factors of cardiovascular risk)
* Previous participation in supervised exercise programs in the last 3 months
* Smoking absence in the last 6 months.

Exclusion Criteria:

* Diagnosis of type 2 diabetes for less than a year
* Glycosylated haemoglobin above 10%
* Pharmacological regimen less than three months
* Main complications of diabetes (diabetic retinopathy, diabetic nephropathy, diabetic foot and main factors of cardiovascular risk)
* Sedentary participants
* Smoking participants

Max Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2023-07-18 (Actual); Study Completion 2023-07-18 (Actual)

PRIMARY OUTCOMES:
Changes from pre- to pos intervention on glycated haemoglobin | Baseline and week 8
  A venous blood sample from the arm will be collected and glycated hemoglobin will be measured and expressed in mmol/mol and as a percentage (%).

SECONDARY OUTCOMES:
Changes from pre- to post intervention in insulin resistance index and β-cell capacity | Baseline and week 8
  A venous blood sample from the arm will be collected and fasting blood glucose (mg/dL) and fasting blood insulin (micro international unit/dL) will be measured, which will determine the homeostasis model assessment (mmol/dL) and homeostasis model assessment 2 for β-cell function (%).
Changes from pre- to pos intervention in angiogenesis | Baseline and week 8
  A venous blood sample from the arm will be collected and, serum Hypoxia Inducible Factor 1 alpha (HIF1-α) will be measured using specific ELISA kit instructions.

OTHER OUTCOMES:
Changes from pre- to pos intervention on cardiovascular risk factor | Baseline and week 8
  A venous blood sample from the arm will be collected and C-Reactive Protein will be measured and expressed in mg/L.
Changes from pre- to pos intervention respiratory and pulmonary gas-exchange variables | Baseline and week 8
  Minute ventilation, oxygen uptake, carbon dioxide production and oxygen saturation, in mL/min, will be measured using the new telemetric portable gas analyser K5 (Rome, Italy), which will be connected to the participants through a traditional facemask and will be calibrated according to manufacturing setting.
Changes from pre- to pos intervention on body composition | Baseline and week 8
  Fat mass (FM) and fat-free mass (FFM) were determined by using whole-body dual-energy X-ray absorptiometry (Lunar Prodigy; General Electric Corp.).
Changes from pre- to pos intervention on body mass index (BMI) | Baseline and week 8
  Height (in meters) will be measured with use of a stadiometer (SECA) and weight (in kilograms) will be measured by using whole-body dual-energy X-ray absorptiometry (Lunar Prodigy; General Electric Corp.), which will determine the BMI, in kg/m^2.
Changes from pre- to pos intervention on waist circumference | Baseline and week 8
  Waist circumference will be measured by using a tape measure (centimeters) positioned 3 centimeters above the iliac crest.
Changes from pre- to pos intervention on blood pressure | Baseline and week 8
  Systolic, diastolic, and mean blood pressure will be measured using an automated sphygmomanometer (Dinamap Pro; Medical Systems, Tampa, FL).
Changes from pre- to pos intervention on lipid profile | Baseline and week 8
  A venous blood sample from the arm will be collected and total cholesterol, LDL cholesterol, HDL cholesterol and triglycerides will be measured and expressed mg/dL.

CONTACTS AND LOCATIONS:
Locations (2):
- Portugal (2):
  - University of Porto, Porto
  - University of Maia, Porto

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Evert AB, Boucher JL, Cypress M, Dunbar SA, Franz MJ, Mayer-Davis EJ, Neumiller JJ, Nwankwo R, Verdi CL, Urbanski P, Yancy WS Jr. Nutrition therapy recommendations for the management of adults with diabetes. Diabetes Care. 2014 Jan;37 Suppl 1:S120-43. doi: 10.2337/dc14-S120. No abstract available. PMID 24357208
- [Background] Miyashita Y, Koide N, Ohtsuka M, Ozaki H, Itoh Y, Oyama T, Uetake T, Ariga K, Shirai K. Beneficial effect of low carbohydrate in low calorie diets on visceral fat reduction in type 2 diabetic patients with obesity. Diabetes Res Clin Pract. 2004 Sep;65(3):235-41. doi: 10.1016/j.diabres.2004.01.008. PMID 15331203
- [Background] Elhayany A, Lustman A, Abel R, Attal-Singer J, Vinker S. A low carbohydrate Mediterranean diet improves cardiovascular risk factors and diabetes control among overweight patients with type 2 diabetes mellitus: a 1-year prospective randomized intervention study. Diabetes Obes Metab. 2010 Mar;12(3):204-9. doi: 10.1111/j.1463-1326.2009.01151.x. PMID 20151996
- [Background] Davis NJ, Tomuta N, Schechter C, Isasi CR, Segal-Isaacson CJ, Stein D, Zonszein J, Wylie-Rosett J. Comparative study of the effects of a 1-year dietary intervention of a low-carbohydrate diet versus a low-fat diet on weight and glycemic control in type 2 diabetes. Diabetes Care. 2009 Jul;32(7):1147-52. doi: 10.2337/dc08-2108. Epub 2009 Apr 14. PMID 19366978
- [Background] Kirk JK, Graves DE, Craven TE, Lipkin EW, Austin M, Margolis KL. Restricted-carbohydrate diets in patients with type 2 diabetes: a meta-analysis. J Am Diet Assoc. 2008 Jan;108(1):91-100. doi: 10.1016/j.jada.2007.10.003. PMID 18155993
- [Background] Millet GP, Debevec T, Brocherie F, Malatesta D, Girard O. Therapeutic Use of Exercising in Hypoxia: Promises and Limitations. Front Physiol. 2016 Jun 10;7:224. doi: 10.3389/fphys.2016.00224. eCollection 2016. No abstract available. PMID 27375500
- [Background] Haider T, Casucci G, Linser T, Faulhaber M, Gatterer H, Ott G, Linser A, Ehrenbourg I, Tkatchouk E, Burtscher M, Bernardi L. Interval hypoxic training improves autonomic cardiovascular and respiratory control in patients with mild chronic obstructive pulmonary disease. J Hypertens. 2009 Aug;27(8):1648-54. doi: 10.1097/HJH.0b013e32832c0018. PMID 19387363
- [Background] Burtscher M, Pachinger O, Ehrenbourg I, Mitterbauer G, Faulhaber M, Puhringer R, Tkatchouk E. Intermittent hypoxia increases exercise tolerance in elderly men with and without coronary artery disease. Int J Cardiol. 2004 Aug;96(2):247-54. doi: 10.1016/j.ijcard.2003.07.021. PMID 15262041
- [Background] Urdampilleta A, Gonzalez-Muniesa P, Portillo MP, Martinez JA. Usefulness of combining intermittent hypoxia and physical exercise in the treatment of obesity. J Physiol Biochem. 2012 Jun;68(2):289-304. doi: 10.1007/s13105-011-0115-1. Epub 2011 Nov 3. PMID 22045452
- [Background] Faramoushi M, Amir Sasan R, Sari Sarraf V, Karimi P. Cardiac fibrosis and down regulation of GLUT4 in experimental diabetic cardiomyopathy are ameliorated by chronic exposures to intermittent altitude. J Cardiovasc Thorac Res. 2016;8(1):26-33. doi: 10.15171/jcvtr.2016.05. Epub 2016 Mar 14. PMID 27069564
- [Background] Little JP, Gillen JB, Percival ME, Safdar A, Tarnopolsky MA, Punthakee Z, Jung ME, Gibala MJ. Low-volume high-intensity interval training reduces hyperglycemia and increases muscle mitochondrial capacity in patients with type 2 diabetes. J Appl Physiol (1985). 2011 Dec;111(6):1554-60. doi: 10.1152/japplphysiol.00921.2011. Epub 2011 Aug 25. PMID 21868679
- [Background] Wolever TM. Carbohydrate and the regulation of blood glucose and metabolism. Nutr Rev. 2003 May;61(5 Pt 2):S40-8. doi: 10.1301/nr.2003.may.S40-S48. PMID 12828191
- [Background] Sousa A, Figueiredo P, Zamparo P, Pyne DB, Vilas-Boas JP, Fernandes RJ. Exercise Modality Effect on Bioenergetical Performance at V O2max Intensity. Med Sci Sports Exerc. 2015 Aug;47(8):1705-13. doi: 10.1249/MSS.0000000000000580. PMID 25412298
- [Derived] Kindlovits R, Sousa AC, Viana JL, Milheiro J, Oliveira BMPM, Marques F, Santos A, Teixeira VH. Evaluating the Therapeutic Potential of Exercise in Hypoxia and Low-Carbohydrate, High-Fat Diet in Managing Hypertension in Elderly Type 2 Diabetes Patients: A Novel Intervention Approach. Nutrients. 2025 Jan 30;17(3):522. doi: 10.3390/nu17030522. PMID 39940380